CLINICAL TRIAL: NCT06847490
Title: Development and Validation of a Predictive Model for Transfusion in Major Abdominal Surgery
Brief Title: Transfusion Prediction in Major Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Ji-Hoon Sim, Assistant Professor, Asan Medical Center
Other Study IDs: AMC (2024-1087)
Record Dates: First submitted 2025-02-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Transfusions
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | US Export: No

INTERVENTIONS:
Other: No intervention (observational study) — This is an observational study aimed at developing and validating a predictive model for perioperative blood transfusion. The study utilizes retrospective clinical data from surgical patients to identify key risk factors associated with transfusion requirements. No experimental intervention will be applied to participants, as the study solely focuses on data analysis and model development.

SUMMARY:
The transfusion nomogram, integrating preoperative variables, may effectively predict intraoperative transfusion in major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older who underwent major abdominal surgery

Exclusion Criteria:

* Patients with known hematologic disease or coagulopathy
* Patients who received a blood transfusion before surgery
* Patients with incomplete data or missing laboratory values

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients (≥18 years old) who underwent major abdominal surgery at a tertiary medical center. The study population consists of patients with available preoperative clinical and laboratory data, allowing for the development of a predictive model for intraoperative blood transfusion. Patients with known hematologic disorders, coagulopathy, or prior transfusion before surgery are excluded to minimize confounding factors.
Sampling Method: Non-Probability Sample
Enrollment: 128749 (Actual)
Dates: Start 2024-06-30 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
Intraoperative transfusion | From surgical incision to the end of surgery
  The primary outcome measure is the occurrence of intraoperative blood transfusion. This includes any administration of red blood cells, plasma, or platelets during the surgical procedure. The study aims to predict transfusion requirements based on preoperative clinical factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, Songpa, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sim JH, Oh AR, Kim S, Park YS, Ha S, Kim JU. Development and validation of a predictive model for transfusion in major abdominal surgery: a multicentre retrospective study. Br J Anaesth. 2025 Sep;135(3):623-631. doi: 10.1016/j.bja.2025.05.048. Epub 2025 Jul 18. PMID 40681389